CLINICAL TRIAL: NCT05997264
Title: A Randomized, Double-blinded, Multicenter Study in Healthy Adults to Evaluate Safety and Immunogenicity of AV7909 Administered at Two Dose Levels on Two Vaccination Schedules, Including a Primary Series and Booster Doses
Brief Title: Anthrax AV7909 Boost Evaluation Study
Acronym: ABESt
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Collaborators: Rho Federal Systems Division, Inc. (Industry); ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ABST001
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Anthrax
MeSH Terms: conditions — Anthrax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Full Dose Schedule 1 (Experimental): This study group will receive full dose AV7909 (0.5mL) at study days 1, 15, 181 and 366. A placebo full dose (0.5 mL) will be administered between the second and third dose of AV7909 at study day 29.
  Update: Enrollment to this treatment arm was closed on 13 May 2024.
  Interventions: Biological: AV7909 Full Dose (0.5 mL)
- Full Dose Schedule 2 (Experimental): This study group will receive of AV7909 full dose (0.5 mL) at study days 1, 29, 181 and 366. A placebo full dose (0.5 mL) will be administered between the first and second dose of AV7909 at study day 15.
  Update: Enrollment to this treatment arm was closed on 13 May 2024.
  Interventions: Biological: AV7909 Full Dose (0.5 mL)
- Half Dose Schedule 1 (Experimental): This study group will receive of AV7909 half dose (0.25 mL) at study days 1, 15, 181 and 366. A placebo half dose (0.25 mL) will be administered between the second and third dose of AV7909 at study day 29.
  Interventions: Biological: AV7909 Half Dose (0.25 mL)
- Half Dose Schedule 2 (Experimental): This study group will receive of AV7909 half dose (0.25 mL) at study days 1, 29, 181 and 366. A placebo full dose (0.25 mL) will be administered between the first and second dose of AV7909 at study day 15.
  Interventions: Biological: AV7909 Half Dose (0.25 mL)

INTERVENTIONS:
Biological: AV7909 Full Dose (0.5 mL) — AV7909 Anthrax Vaccine is being developed by Emergent Product Development Gaithersburg Inc. (Emergent) for PEP of disease in persons 18 through 65 years of age following suspected or confirmed B. anthracis exposure when administered in conjunction with the recommended antibacterial regimen. AV7909 is a combination product containing BioThrax and CPG 7909, a synthetic immunostimulatory oligodeoxynucleotide that has been shown to be a potent vaccine adjuvant. CPG 7909 is a Toll-like receptor 9 agonist designed to induce both an enhanced antigen-specific antibody response and a natural killer T-cell immune response when used in combination with prophylactic (preventative) or therapeutic vaccines.
  Arms: Full Dose Schedule 1; Full Dose Schedule 2
Biological: AV7909 Half Dose (0.25 mL) — AV7909 Anthrax Vaccine is being developed by Emergent Product Development Gaithersburg Inc. (Emergent) for PEP of disease in persons 18 through 65 years of age following suspected or confirmed B. anthracis exposure when administered in conjunction with the recommended antibacterial regimen. AV7909 is a combination product containing BioThrax and CPG 7909, a synthetic immunostimulatory oligodeoxynucleotide that has been shown to be a potent vaccine adjuvant. CPG 7909 is a Toll-like receptor 9 agonist designed to induce both an enhanced antigen-specific antibody response and a natural killer T-cell immune response when used in combination with prophylactic (preventative) or therapeutic vaccines.
  Arms: Half Dose Schedule 1; Half Dose Schedule 2

SUMMARY:
This randomized, phase 2, double-blinded, multicenter study is designed to assess the safety and immune response kinetics of CYFENDUS™ (henceforth AV7909) administered on 2 primary series vaccination schedules followed by 6- and 12-month boosters.

DETAILED DESCRIPTION:
This trial is a randomized, double-blinded, multicenter study designed to evaluate safety and immune response kinetics of full and half doses of AV7909 administered on 2 primary series vaccination schedules followed by 6- and 12-month boosters. Healthy adult male and female subjects aged 18 through 65 years, inclusive, will be screened for baseline health status to ensure trial eligibility. Subjects meeting all the inclusion and none of the exclusion criteria will be randomized to receive either half or full doses of AV7909 on 1 of 2 vaccination schedules. Randomization will be stratified by sex. Subjects will be randomized 1:1:1:1 within stratum across 4 treatment groups (approximately 55 subjects per group). Subjects will receive a total of 5 intramuscular (IM) injections. Primary series IP doses will be administered on Days 1, 15, and 29, and booster IP doses will be administered on Days 181 and 366. On each IP administration day, each subject will receive an IM injection of full-dose AV7909 (0.5 mL), half-dose AV7909 (0.25 mL), or placebo (0.5 mL or 0.25 mL sodium chloride for injection), based on their assigned treatment group.

Update: The 2 treatment groups (Study Groups 1 and 2) in which subjects are to receive full doses of AV7909 were closed to enrollment on 13 May 2024 to preserve resources for the groups that BARDA considers the highest priority and reflects no concerns due to a safety signal or request of the Data Safety Monitoring Board (DSMB). Subjects randomized prior to this date will continue in the study in their assigned treatment group as described in the protocol. Subjects randomized on or after 13 May 2024 will be randomized 1:1 within stratum across the 2 remaining treatment groups (Study Groups 3 and 4), and on each IP administration day will receive an IM injection of half-dose AV7909 (0.25 mL) or placebo (0.25 mL sodium chloride for injection), based on their assigned treatment group. There are no other changes to the study protocol.

Safety assessments will be based on solicited adverse events (AEs; local and systemic reactogenicity symptoms) with onset within 7 days after each IP administration; unsolicited treatment-emergent adverse events (TEAEs) with onset within 30 days after each IP administration; and treatment-emergent serious adverse events (SAEs), potentially immune-mediated medical conditions (PIMMCs), and medically attended adverse events (MAAEs) occurring during study participation (ie, up to 1 year after the last IP administration). For this study, a PIMMC is considered to be unexpected and will be treated as a serious and unexpected suspected adverse reaction (SUSAR) per 21 CFR 312.32.

Immunogenicity assessments will include geometric mean titer (GMT), seroprotection rate, and seroconversion rate by toxin-neutralizing antibody (TNA) 50% neutralization factor (NF50) and enzyme-linked immunosorbent assay (ELISA) anti-protective antigen (PA) Immunoglobulin G (IgG).

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant females, 18 through 65 years of age, inclusive.
2. Willing and able to provide written informed consent prior to initiation of study procedures.
3. In relatively stable health, as determined by medical history and physical examination. Any chronic medical diagnoses or conditions should be stable and well managed, with no significant changes expected during the study period, and in the opinion of the site investigator, will not impact the ability to assess safety and/or immunogenicity per the study design.
4. If a female of childbearing potential who is sexually active, agrees to use an acceptable method of birth control from Screening to Day 396 and has used a reliable birth control method for at least 2 months prior to Screening.

   1. Female of childbearing potential is defined as post onset menarche and pre-menopausal person capable of becoming pregnant. This does not include females who meet any of the following conditions: a) menopausal >2 years; b) tubal ligation >1 year; c) bilateral salpingo-oophorectomy; or d) hysterectomy.
   2. Adequate contraception is defined as a contraceptive method with a failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label, for example: oral contraceptives, either combined or progestogen alone; injectable progestogen; implants of etenogestrel or levonorgestrel; estrogenic vaginal ring; percutaneous contraceptive patches; intrauterine device or intrauterine system; the female subject has exclusively female sexual partners; partner is sterile or otherwise unable to produce sperm (information on the person's sterility can come from the site personnel's review of the subject's medical records or interview with the subject regarding her medical history); male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository); or male condom combined with a female diaphragm, either with or without a vaginal spermicide (foam, gel, film, cream, or suppository).
5. Available for all study visits, willing to participate in all study procedures, and not planning to relocate from the area for the duration of the study.
6. Has a body mass index (BMI) greater than 18.0 and less than 35.0 kg/m2, inclusive

Exclusion Criteria:

1. Has an acute illness, as determined by the site investigator, within 72 hours prior to study IP administration.

   * An acute illness that is nearly resolved, with only minor residual symptoms remaining, is allowable if, in the opinion of the site investigator, the residual symptoms will not interfere with the ability of study staff to assess safety parameters as required by the protocol.
   * If the subject's temperature is above 100.4°F, indicating illness, the subject may be re-assessed for eligibility a minimum of 24 hours later.
2. Has a history of severe reactions to components of AV7909.
3. Has a history of anthrax disease, suspected exposure to anthrax, or previous vaccination with any anthrax vaccine.
4. Has recently diagnosed or poorly controlled human immunodeficiency virus (HIV).
5. Has an acute or chronic hepatitis B or hepatitis C infection, as identified through laboratory testing.

   - A subject who has been effectively treated for hepatitis C, as evidenced by a negative hepatitis C ribonucleic acid (RNA) confirmation test, and who no longer requires antiviral therapy is not excluded.
6. Is suffering from or has a history of neuralgia, paresthesia, neuritis, convulsions, or encephalomyelitis within 90 days prior to Screening, or a family history of Guillain-Barré syndrome.
7. Has a history of alcohol or drug abuse within 5 years prior to Screening.
8. Has any diagnosis, current or past, of schizophrenia, bipolar disease, or any other psychiatric diagnosis that may, in the opinion of the site investigator, interfere with subject compliance or safety evaluations.
9. Is taking herbal medicines/preparations that are known to have a direct or indirect effect on the immune system.
10. Presence of tattoos on both upper arms that would cover or partially cover all potential vaccination sites.
11. Clinically relevant signs of pathology or conduction disturbances documented by electrocardiogram (EKG).
12. Has taken corticosteroids as follows within 30 days prior to Screening.

    * Oral or parenteral corticosteroids at a dose of ≥20 mg daily and/or
    * High-dose (>800 mcg/day of beclomethasone di-iso-propionate chlorofluorocarbon [CFC] or equivalent) inhaled corticosteroids.
13. Female of childbearing potential who has a positive urine pregnancy test or who is currently breastfeeding.
14. Has had any vaccination (licensed or under Emergency Use Authorization [EUA]; any type) within the 30 days prior to the planned first study IP administration.
15. Is immunosuppressed due to an underlying disease or medication, use of anticancer chemotherapy (cytotoxic), or radiation therapy.
16. With the exception of basal or squamous cell skin cancer, has known active neoplastic disease, including hematologic malignancy.
17. Has received an investigational agent within 30 days prior to the planned first study IP administration.
18. Has any laboratory test result or clinical findings (including vital signs) that singly or in combination are likely to unfavorably alter the risks of subject participation or to confound study safety or immunogenicity results, in the opinion of the site investigator. Additionally, the following are exclusionary:

    1. Has any clinically significant Grade 3 laboratory or vital sign result, or any Grade 4 laboratory or vital sign result (regardless of assessed significance) at Screening.
    2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 times the upper limit of normal (ULN), or bilirubin >1.5 times the ULN unless isolated Gilbert's syndrome.
    3. Creatinine >1.5 times ULN for age and sex.
    4. White blood cell count <3,000/µL or >12,500/µL; absolute neutrophil count <1,200/µL; absolute lymphocyte count <750/µL; hemoglobin <10 g/dL females, or <11.5 g/dL males; platelet count <75,000/µL.
    5. Hemoglobin A1c (HbA1c) >7.0% at Screening.
19. Has any disease or medical condition that, in the opinion of the site investigator, might confound interpretation of safety or immunogenicity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
All solicited local and systemic reactogenicity symptoms with onset within 7 days after each IP administration day. | Within 7 days after each IP administration.
Geometric mean titer (GMT) as measured by toxin-neutralizing antibody (TNA) 50% neutralization | Day 64

SECONDARY OUTCOMES:
Unsolicited treatment-emergent adverse events (TEAEs) with onset within 30 days after each IP administration day. | Within 30 days after each IP administration.
Treatment-emergent serious adverse events (SAEs) up to 1 year after the last IP administration day. | Within 1 year after the last IP administration.
Treatment-emergent potentially immune-mediated medical conditions (PIMMCs) up to 1 year after the last IP administration day. | Within 1 year after the last IP administration.
Treatment-emergent medically attended adverse events (MAAEs) up to 1 year after the last IP administration day. | Within 1 year after the last IP administration.
Geometric mean titer (GMT) as measured by toxin-neutralizing antibody (TNA) 50% neutralization factor (NF50) at Day 15, Day 29, Day 36, Day 43, Day 50, Day 85, Day 181, Day 211, Day 366, Day 396, Day 546, and Day 731. | Day 15 through 731.
Seroprotection rate as measured by toxin-neutralizing antibody (TNA) 50% neutralization factor (NF50) at Day 15, Day 29, Day 36, Day 43, Day 50, Day 64, Day 85, Day 181, Day 211, Day 366, Day 396, Day 546, and Day 731. | Day 15 through 731.
Geometric mean titer (GMT) as measured by ELISA anti-PA IgG at Day 15, Day 29, Day 36, Day 43, Day 50, Day 64, Day 85, Day 181, Day 211, Day 366, Day 396, Day 546, and Day 731. | Day 15 through 731.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Eisnor, MD, Study Chair — Biomedical Advanced Research and Development Authority
Locations (6):
- United States (6):
  - Accellacare of Hickory, Hickory, North Carolina
  - Accellacare of Salisbury, Salisbury, North Carolina
  - Accellacare of Piedmont, Statesville, North Carolina
  - Accellacare of Winston-Salem, Winston-Salem, North Carolina
  - Accellacare Knoxville, Jefferson City, Tennessee
  - Accellacare Knoxville, Knoxville, Tennessee